CLINICAL TRIAL: NCT04106921
Title: Evaluation of a Mobile Application Tool for Increasing Community Health Worker Home Visit Coverage: A Randomized Controlled Study
Brief Title: Universal Coverage Mode RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ari Johnson, MD (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Medic Mobile (Industry)
Responsible Party: Sponsor-Investigator, Ari Johnson, MD, MD, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 0219-0619
Record Dates: First submitted 2019-09-25; First posted 2019-09-27 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Community Health Workers
Keywords: community health workers; primary health care; mobile applications

STUDY DESIGN:
Intervention Model Description: Difference in differences parallel randomized controlled trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Universal Health Coverage Mode (Experimental): The NGOs Muso and Medic Mobile have partnered to develop Universal Health Coverage Mode, a smartphone app tool that provides visual cues to help CHWs track the quantity of household visits they have conducted at each household in a given month.
  Interventions: Other: Universal Health Coverage Mode
- Work as usual (No Intervention): For the control arm, all households within the CHW's household list in the app will have the same appearance. There will be no visual differentiation between households on the list to indicate the frequency of home visits.

INTERVENTIONS:
Other: Universal Health Coverage Mode — In the intervention arm, the CHW's household list will appear differently within the app in the following ways:
  The CHW will be able to filter and order households by the date of the most recent home visit.
  A color-coded visual icon will display the number of home visits in the past month for each household.
  A red exclamation mark will be displayed for every household that has not reached 2 visits in the past month (default at the start of every month).
  Text displayed below each household showing the date of last visit will turn red if more than 30 days have passed since last visit. When more than 60 days have passed since the most recent visit, the text displayed below each household showing the date of last visit will be changed to "date of last visit is unknown" in red.
  The family profile will also contain the date of last visit, and the visits they have received in that month
  Arms: Universal Health Coverage Mode

SUMMARY:
Community Health Workers that work in collaboration with the NGO Muso Health and the Malian government in both a peri-urban and a rural site in Mali, provide care proactively to the population they form part of.

To work, they use a smartphone application that was developed as a job aid to support task management, panel management and clinical decision support functions. For this study, a tool called "Universal Health Coverage Mode" was designed to be integrated into the CHW application to help Community Health Workers visit every household at least twice per month.

We hypothesize that Community Health Workers (CHWs) assigned to use Universal Health Coverage (UHC) Mode, a mobile application tool, will achieve higher coverage of homes visited (defined as being visited at least two times in a month) than those without this tool.

DETAILED DESCRIPTION:
Community Health Workers participating in the study will be providing care through the Proactive Community Case Management intervention, described in detail elsewhere. Through this package of services, CHWs are required to conduct at least two hours of home visits per day, six days per week, to achieve a goal of at least two home visits per household per month. All CHWs receive monthly individual supervision via a 360 Supervision protocol, described in detail elsewhere, as well as group supervisions weekly (at the Yirimadio site) or twice-monthly (at the Tori site). At the Tori site, households served by each CHW were previously registered via a population census which is updated every year by an independent team of surveyors. Within the Yirimadio site, all households have been registered by the CHW herself to achieve a ratio of approximately 1000 patients per CHW.

CHWs at both sites and both arms of the study will also receive monthly performance feedback via a CHW Performance Dashboard, described elsewhere, which provides personalized feedback on the quantity, speed, and coverage of care. CHW supervisors will be able to see their supervisees' performance data and provide feedback via the monthly supervisions. CHWs at both sites will receive feedback for community care management indicators, but only Yirimadio's CHW supervisors will observe CHWs performance on proactive household visits.

All CHWs at both sites use a CHW App, a free and open source smartphone application developed by Medic Mobile with Muso. The CHW App is a job aid that supports task management, panel management, and clinical decision support functions, while providing a mechanism for data collection and submission. Previously, CHWs had to manage 14 different types of paper forms that their core workflow entails, and the data was entered by hand for each of these forms to carry out monitoring and evaluation tasks. Now, there is no need for photocopying, carrying and stocking all 14 forms, and data is automatically sent to a central database once the smartphones are synchronized. Also, for CHW tracking their patients and the tasks they performed meant a huge organizational challenge. The app was modeled to tackle this problem using a human centered design, allowing the CHWs to easily search for and access their patients registries and histories.

For the control arm, all households within the CHW's household list in the app will have the same appearance. There will be no visual differentiation between households on the list to indicate the frequency of home visits.

In the intervention arm, the CHW's household list will appear differently within the app in the following ways:

The CHW will be able to filter and order households by the date of the most recent home visit, to identify households that have been visited least frequently.

A color-coded visual icon will display the number of home visits in the past month for each household.Red color for 0 home visits for a household in the past month (default at the start of every month).Orange color for 1 home visit for a household in the past month.Blue color for 2 or more visits for a household in the past month.

A red exclamation mark will be displayed for every household that has not reached 2 visits in the past month (default at the start of every month).

Text displayed below each household showing the date of last visit will turn red if more than 30 days have passed since last visit. When more than 60 days have passed since the most recent visit, the text displayed below each household showing the date of last visit will be changed to "date of last visit is unknown" in red.

The family profile will also contain the date of last visit, and the visits they have received in that month.

ELIGIBILITY:
Inclusion Criteria:

* Community Health Workers serving the Tori (n=27) and Yirimadio (n=172) catchment areas conducting proactive home visits will be eligible to participate in the study

Exclusion Criteria:

* CHWs involved in pilot-testing UHC Mode prior to the trial will be excluded from the trial.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-07-26 (Actual); Study Completion 2019-07-26 (Actual)

PRIMARY OUTCOMES:
Primary outcome | 4 months
  The probability of a household receiving two or more visits per "workflow" month (a month being from the 26th of one month to the 25th of the next month).

SECONDARY OUTCOMES:
Secondary outcome 1 | 4 months
  Number of days between household visits for each household served by CHWs
Secondary outcome 2 | 4 months
  Number of visits per household per "workflow"month
Secondary outcome 3 | 4 months
  Percentage of sick individuals in a household visited within 24 hours (among households with a sick person).

CONTACTS AND LOCATIONS:
Locations (1):
- Muso, Bamako, Mali

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] GBD 2015 SDG Collaborators. Measuring the health-related Sustainable Development Goals in 188 countries: a baseline analysis from the Global Burden of Disease Study 2015. Lancet. 2016 Oct 8;388(10053):1813-1850. doi: 10.1016/S0140-6736(16)31467-2. Epub 2016 Sep 21. PMID 27665228
- [Background] Rasanathan K, Muniz M, Bakshi S, Kumar M, Solano A, Kariuki W, George A, Sylla M, Nefdt R, Young M, Diaz T. Community case management of childhood illness in sub-Saharan Africa - findings from a cross-sectional survey on policy and implementation. J Glob Health. 2014 Dec;4(2):020401. doi: 10.7189/jogh.04.020401. PMID 25520791
- [Background] Young M, Wolfheim C, Marsh DR, Hammamy D. World Health Organization/United Nations Children's Fund joint statement on integrated community case management: an equity-focused strategy to improve access to essential treatment services for children. Am J Trop Med Hyg. 2012 Nov;87(5 Suppl):6-10. doi: 10.4269/ajtmh.2012.12-0221. PMID 23136272
- [Background] Black RE, Taylor CE, Arole S, Bang A, Bhutta ZA, Chowdhury AMR, Kirkwood BR, Kureshy N, Lanata CF, Phillips JF, Taylor M, Victora CG, Zhu Z, Perry HB. Comprehensive review of the evidence regarding the effectiveness of community-based primary health care in improving maternal, neonatal and child health: 8. summary and recommendations of the Expert Panel. J Glob Health. 2017 Jun;7(1):010908. doi: 10.7189/jogh.07.010908. PMID 28685046
- [Background] Freeman PA, Schleiff M, Sacks E, Rassekh BM, Gupta S, Perry HB. Comprehensive review of the evidence regarding the effectiveness of community-based primary health care in improving maternal, neonatal and child health: 4. child health findings. J Glob Health. 2017 Jun;7(1):010904. doi: 10.7189/jogh.07.010904. PMID 28685042
- [Background] Jennings MC, Pradhan S, Schleiff M, Sacks E, Freeman PA, Gupta S, Rassekh BM, Perry HB. Comprehensive review of the evidence regarding the effectiveness of community-based primary health care in improving maternal, neonatal and child health: 2. maternal health findings. J Glob Health. 2017 Jun;7(1):010902. doi: 10.7189/jogh.07.010902. PMID 28685040
- [Background] Perry HB, Zulliger R, Rogers MM. Community health workers in low-, middle-, and high-income countries: an overview of their history, recent evolution, and current effectiveness. Annu Rev Public Health. 2014;35:399-421. doi: 10.1146/annurev-publhealth-032013-182354. Epub 2014 Jan 2. PMID 24387091
- [Background] Sacks E, Freeman PA, Sakyi K, Jennings MC, Rassekh BM, Gupta S, Perry HB. Comprehensive review of the evidence regarding the effectiveness of community-based primary health care in improving maternal, neonatal and child health: 3. neonatal health findings. J Glob Health. 2017 Jun;7(1):010903. doi: 10.7189/jogh.07.010903. PMID 28685041
- [Background] Munos M, Guiella G, Roberton T, Maiga A, Tiendrebeogo A, Tam Y, Bryce J, Baya B. Independent Evaluation of the Rapid Scale-Up Program to Reduce Under-Five Mortality in Burkina Faso. Am J Trop Med Hyg. 2016 Mar;94(3):584-595. doi: 10.4269/ajtmh.15-0585. Epub 2016 Jan 19. PMID 26787147
- [Background] Amouzou A, Kanyuka M, Hazel E, Heidkamp R, Marsh A, Mleme T, Munthali S, Park L, Banda B, Moulton LH, Black RE, Hill K, Perin J, Victora CG, Bryce J. Independent Evaluation of the Integrated Community Case Management of Childhood Illness Strategy in Malawi Using a National Evaluation Platform Design. Am J Trop Med Hyg. 2016 Jun 1;94(6):1434-1435. doi: 10.4269/ajtmh.16-0110b. No abstract available. PMID 27252480
- [Background] Amouzou A, Hazel E, Shaw B, Miller NP, Tafesse M, Mekonnen Y, Moulton LH, Bryce J, Black RE. Effects of the integrated Community Case Management of Childhood Illness Strategy on Child Mortality in Ethiopia: A Cluster Randomized Trial. Am J Trop Med Hyg. 2016 Mar;94(3):596-604. doi: 10.4269/ajtmh.15-0586. Epub 2016 Jan 19. PMID 26787148
- [Background] Hazel E, Bryce J, The Iip-Jhu iCCM Evaluation Working Group. On Bathwater, Babies, and Designing Programs for Impact: Evaluations of the Integrated Community Case Management Strategy in Burkina Faso, Ethiopia, and Malawi. Am J Trop Med Hyg. 2016 Mar;94(3):568-570. doi: 10.4269/ajtmh.94-3intro1. No abstract available. PMID 26936991
- [Background] Johnson A, Goss A, Beckerman J, Castro A. Hidden costs: the direct and indirect impact of user fees on access to malaria treatment and primary care in Mali. Soc Sci Med. 2012 Nov;75(10):1786-92. doi: 10.1016/j.socscimed.2012.07.015. Epub 2012 Aug 1. PMID 22883255
- [Background] Johnson AD, Thiero O, Whidden C, Poudiougou B, Diakite D, Traore F, Samake S, Kone D, Cisse I, Kayentao K. Proactive community case management and child survival in periurban Mali. BMJ Glob Health. 2018 Mar 12;3(2):e000634. doi: 10.1136/bmjgh-2017-000634. eCollection 2018. PMID 29607100
- [Background] Linn AM, Ndiaye Y, Hennessee I, Gaye S, Linn P, Nordstrom K, McLaughlin M. Reduction in symptomatic malaria prevalence through proactive community treatment in rural Senegal. Trop Med Int Health. 2015 Nov;20(11):1438-1446. doi: 10.1111/tmi.12564. Epub 2015 Aug 7. PMID 26171642
- [Background] Johnson AD, Thomson DR, Atwood S, Alley I, Beckerman JL, Kone I, Diakite D, Diallo H, Traore B, Traore K, Farmer PE, Murray M, Mukherjee J. Assessing early access to care and child survival during a health system strengthening intervention in Mali: a repeated cross sectional survey. PLoS One. 2013 Dec 11;8(12):e81304. doi: 10.1371/journal.pone.0081304. eCollection 2013. PMID 24349053
- [Background] Whidden C, Kayentao K, Liu JX, Lee S, Keita Y, Diakite D, Keita A, Diarra S, Edwards J, Yembrick A, Holeman I, Samake S, Plea B, Coumare M, Johnson AD. Improving Community Health Worker performance by using a personalised feedback dashboard for supervision: a randomised controlled trial. J Glob Health. 2018 Dec;8(2):020418. doi: 10.7189/jogh.08.020418. PMID 30333922
- [Derived] Yang JE, Lassala D, Liu JX, Whidden C, Holeman I, Keita Y, Djiguiba Y, N'Diaye SI, Fall F, Kayentao K, Johnson AD. Effect of mobile application user interface improvements on minimum expected home visit coverage by community health workers in Mali: a randomised controlled trial. BMJ Glob Health. 2021 Nov;6(11):e007205. doi: 10.1136/bmjgh-2021-007205. PMID 34815242